CLINICAL TRIAL: NCT03792438
Title: Study of the Vascularity of Uterine Septum Using Three Dimensional Power Doppler Ultrasound
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Mohamed Elnaggar, Principal Investigator, Ain Shams Maternity Hospital
Other Study IDs: Hesham Mohamed Elnaggar
Record Dates: First submitted 2018-12-26; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Septum; Uterus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transvaginal 3D Power Doppler Ultrasound — Samsung H60 ultrasound machine with 4-9 MHz volume transducer using VOCAL system and Histogram Facility

SUMMARY:
This study aims to assess the relation between the vascularity of uterine septum and obstetric performance with Transvaginal 3D Power Doppler Ultrasound

DETAILED DESCRIPTION:
Research hypothesis:

In women with uterine septum vascularity of the septum may affect obstetric performance.

Research question:

In women with uterine septum does vascularity of the septum affect obstetric outcome?

ELIGIBILITY:
Inclusion Criteria:

* Patients with septate uterus diagnosed by office hysteroscopy

Exclusion Criteria:

* Women with previous uterine scar.
* Women with suspected or confirmed pregnancy.
* Women with active pelvic infection or old one.
* Women with abnormal uterine bleeding.
* Fibroids, adenomyosis or ovarian swelling.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Patients with primary infertility or recurrent abortion attending to Early Cancer Detection Unit at Ain Shams Maternity Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-05-27 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with high vascular indices (VI, FI, VFI) in relation to Vascular indices of the rest of the surrounding myometrium | About 18 months
  Number of participants with high vascular indices (VI, FI, VFI) in relation to Vascular indices of the rest of the surrounding myometrium and its relationship to either primary infertility or recurrent abortion

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Amer, MD, Study Chair — Professor; Nashwa E Hassan, MD, Study Director — Assistant Professor; Mortada E Ahmed, MD, Study Director — Lecturer
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No